CLINICAL TRIAL: NCT00617461
Title: Study PXN110527: The Investigation of the Efficacy and Pharmacokinetics of XP13512 in Subjects With Neuropathic Pain Associated With Post-herpetic Neuralgia (PHN) Who Have Had an Inadequate Response to Gabapentin Treatment.
Brief Title: A Clinical Study in Subjects With Neuropathic Pain From PHN Who Have Had an Inadequate Response to Gabapentin Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 110527
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Results first posted 2011-05-20 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-01

CONDITIONS: Neuralgia, Postherpetic
Keywords: Post-herpetic neuralgia(PHN); Neuropathic pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GEn 1200mg/day (Experimental): gabapentin enacarbil 1200mg/day, 4 weeks treatment in either the first or second treatment period
  Interventions: Drug: GEn 1200mg/day
- GEn 3600mg/day (Experimental): gabapentin enacarbil 3600mg/day, 4 weeks treatment in either the first or second treatment period
  Interventions: Drug: GEn 3600mg/day

INTERVENTIONS:
Drug: GEn 1200mg/day — 1200mg/day gabapentin enacarbil
  Other Names: GEn; XP13512/GSK1838262; gabapentin enacarbil
  Arms: GEn 1200mg/day
Drug: GEn 3600mg/day — 3600mg/day gabapentin enacarbil
  Other Names: gabapentin enacarbil; GEn; XP13512/GSK1838262
  Arms: GEn 3600mg/day

SUMMARY:
The purpose of this study is evaluate the difference between two doses of gabapentin enacarbil (XP13512/GSK1838262), hereafter referred to as GEn, on pain associated with post-herpetic neuralgia.

DETAILED DESCRIPTION:
The primary purpose of study PXN110527 was to investigate the efficacy of a high (3600mg/day) dose versus a low (1200mg/day) dose of GEn in subjects with post-herpetic neuralgia (PHN) who have a history of an inadequate response to gabapentin treatment. The study is a cross-over design. Prior to screening subjects are required to have a demonstrated history of an inadequate response (as determined by the investigator) to at least 1800 mg/day of gabapentin. Prior history of treatment with gabapentin includes current treatment at 1800mg/day (2 weeks) or prior treatment with ≥1800mg/day (4 weeks). Subjects could also have been treated with pregabalin monotherapy (150-300mg/day, ≥4 weeks) and had an inadequate response.

Subjects are treated with gabapentin 1800mg/day during the Baseline Period and are randomized if during the Basleline Period they are compliant with gabapentin treatment and have a 24-hour average pain intensity score ≥4.0 based on an 11-point pain intensity numerical rating scale (PI-NRS). Subjects are then randomized to receive gabapentin enacarbil (either 1200mg/day or 3600mg/day in a 1:1 ratio) for Treatment Period 1 (28 days). Followed by a dose of 2400mg/day for 4 days and the alternate fixed dose (either 3600 mg/day or 1200 mg/day) for Treatment Period 2 (28 days).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Documented medical diagnosis of PHN with pain present for at least 3 months from the healing of a herpes zoster rash
* Female subjects are eligible if of non-childbearing potential or not lactating, has a negative pregnancy, and agrees to use one a specified highly effective method for avoiding pregnancy.
* Currently on a stable dose of 1800 mg/day of gabapentin for ≥2 weeks with inadequate response OR
* Not currently treated with gabapentin, but previously treated with ≥1800 mg/day of gabapentin for 4 weeks or more with inadequate response.
* Baseline 24-hour average pain intensity score ≥ 4.0 based on an 11-point PI-NRS
* Provides written informed consent in accordance with all applicable regulatory requirements

Exclusion Criteria:

* Other chronic pain conditions not associated with PHN. However, the subject will not be excluded if:
* The pain is located at a different region of the body; and
* The pain intensity is not greater than the pain intensity of the PHN; and
* The subject can assess PHN pain independently of other pain
* Is unable to discontinue prohibited medications or non-drug therapies or procedures throughout the duration of the study
* Hepatic impairment defined as ALT or AST > 2x upper limit of normal (ULN), or alkaline phosphatase or bilirubin > 1.5x ULN
* Chronic hepatitis B or C
* Impaired renal function defined as creatinine clearance <60 mL/min or requiring hemodialysis
* Corrected QT (QTc) interval ≥ 450 msec or QTc interval ≥480 msec for patients with Bundle Branch Block
* Uncontrolled hypertension at screen (sitting systolic >160 mmHg and/or sitting diastolic >90 mmHg)
* Current diagnosis of active epilepsy or any active seizure disorder requiring chronic therapy with antiepileptic drugs
* Medical condition or disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of GEn, or, in the investigator's judgment
* Is considered to be clinically significant and may pose a safety concern, or,
* Could interfere with the accurate assessment of safety or efficacy, or,
* Could potentially affect a subject's safety or study outcome
* Current or chronic history of liver disease (including acute viral hepatitis), or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Meets criteria defined by the DSM-IV-TR for a major depressive episode or for active significant psychiatric disorders within last year
* Depression in remission, with or without antidepressant treatment, may participate, unless stable antidepressant regimen is a prohibited medication
* Antidepressant medication may not be changed or discontinued to meet entry criteria and must be stable for at least three months prior to enrollment
* History of clinically significant drug or alcohol abuse (DSM-IV-TR) or is unable to refrain from substance abuse throughout the study. Benzodiazepines or atypical benzodiazepines as hypnotic sleep agents permitted.
* Currently participating in another clinical study in which the subject is, or will be exposed to an investigational or non-investigational drug or device
* Has participated in a clinical study and was exposed to investigational or non-investigational drug or device:
* Within preceding month for studies unrelated to PHN, or
* Within preceding six months for studies related to PHN
* Treated previously with GEn
* History of allergic or medically significant adverse reaction to investigational products (including gabapentin) or their excipients, acetaminophen or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (39):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Chipley, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Marianna, Florida
  - GSK Investigational Site, Miami Springs, Florida
  - GSK Investigational Site, Naranja, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Norman, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Greensburg, Pennsylvania
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Yakima, Washington
- Germany (10):
  - GSK Investigational Site, Schönau, Baden-Wurttemberg
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Berlin, State of Berlin

REFERENCES:
- [Derived] Harden RN, Freeman R, Rainka M, Zhang L, Bell C, Berges A, Chen C, Graff O, Harding K, Hunter S, Kavanagh S, Schwartzbach C, Warren S, McClung C. A phase 2a, randomized, crossover trial of gabapentin enacarbil for the treatment of postherpetic neuralgia in gabapentin inadequate responders. Pain Med. 2013 Dec;14(12):1918-32. doi: 10.1111/pme.12227. Epub 2013 Sep 18. PMID 24102928

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) were enrolled in a two-week Baseline Period, which included treatment with 1800 milligrams (mg)/day gabapentin. Participants who met entry criteria were then randomized. Inv., investigator.
Groups:
- GEn 1200 mg/Day Followed by GEn 3600 mg/Day: Gabapentin enacarbil (XP13512/GSK1838262), hereafter referred to as GEn, 1200 mg/day administered for 28 days, followed by a 4-day crossover period during which participants received GEn 2400 mg/day. After the crossover period, participants switched to a dose of 3600 mg/day for 28 days. After completion of the second treatment period, participants entered a down-titration period in which they received 1200 mg/day for 3 days, followed by 600 mg/ day for 3 days.
- GEn 3600 mg/Day Followed by GEn 1200 mg/Day: GEn 3600 mg/day administered for 28 days, followed by a 4-day crossover period during which participants received GEn 2400 mg/day. After the crossover period, participants switched to a dose of 1200 mg/day for 28 days. After completion of the second treatment period, participants entered a down-titration period in which they received 2400 mg/day for 2 days, followed by 1200 mg/day for 2 days, followed by 600 mg/day for 2 days.
Period: First Treatment Intervention Period
Arm/Group | GEn 1200 mg/Day Followed by GEn 3600 mg/Day | GEn 3600 mg/Day Followed by GEn 1200 mg/Day
Started | 52 (2 par. (1 withdrawal due to inv. discretion, 1 withdrawal by subject) did not take study drug.) | 44
Completed | 42 | 41
Not Completed | 10 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Investigator Discretion | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0
Period: 4-Day Crossover Period
Arm/Group | GEn 1200 mg/Day Followed by GEn 3600 mg/Day | GEn 3600 mg/Day Followed by GEn 1200 mg/Day
Started | 42 | 40 (One 3600:1200 participant skipped the Crossover period, going directly to second Treatment Period.)
Completed | 41 | 40
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Treatment Intervention Period
Arm/Group | GEn 1200 mg/Day Followed by GEn 3600 mg/Day | GEn 3600 mg/Day Followed by GEn 1200 mg/Day
Started | 41 | 41
Completed | 41 | 37
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 3
Period: 6-Day Down-Titration Period
Arm/Group | GEn 1200 mg/Day Followed by GEn 3600 mg/Day | GEn 3600 mg/Day Followed by GEn 1200 mg/Day
Started | 41 | 37
Completed | 39 | 35
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Did Not Attend Down-titration Visit | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants in the Intent-to-Treat Population: All randomized participants who took at least one dose of study drug and had at least one post-baseline efficacy assessment, summarized independent of treatment sequence.
Arm/Group | All Participants in the Intent-to-Treat Population
Number analyzed (Participants) | 93
Age Continuous [Mean (Standard Deviation); unit: Years] — Age (years) data were collected for all participants at the beginning of the Baseline period. Participants were not included in the Intent-to-Treat (ITT) Population unless they had an average baseline pain rating of 4, were randomized, took at least one dose of investigational product and completed one post-baseline efficacy assessment.
  Years | 63 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender data were collected for all participants at the beginning of the Baseline period. Participants were not included in the Intent-to-Treat (ITT) Population unless they had an average baseline pain rating of 4, were randomized, took at least one dose of investigational product and completed one post-baseline efficacy assessment.
  Participants
    Female | 36
    Male | 57
Race/Ethnicity, Customized [Number; unit: participants] — Race data were collected for all participants at the beginning of the Baseline period. Participants were not included in the Intent-to-Treat (ITT) Population unless they had an average baseline pain rating of 4, were randomized, took at least one dose of investigational product and completed one post-baseline efficacy assessment.
  participants
    African American/African Heritage | 18
    White | 74
    American Indian or Alaska Native & White | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean 24-hour Average Pain Intensity (API) Score at the Last Week of Each Treatment Period Using Last Observation Carried Forward (LOCF) Data
Description: Baseline and end of treatment values are the calculated means of the daily 24-hour API scores for each participant during the last 7 days prior to randomization (baseline) and the last 7 days on treatment within each period (end of treatment). Participants rated their API over the preceding 24 hours, using an 11-point PI-Numerical Rating Scale (0=no pain, 10=pain as bad as you can imagine). LOCF was used if less than 4 days of diary data were provided. Change from baseline was calculated as end of treatment minus baseline. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, 1 participant did not provide post-baseline data for 24-hour API assessments during the GEn 3600mg treatment period, and was therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Groups:
- GEn 1200 mg: GEn 1200 mg daily either in first intervention period or second intervention period
- GEn 3600 mg: GEn 3600 mg daily either in first intervention period or second intervention period
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 90 | 84
points on a scale | -1.18 (0.171) | -1.47 (0.173)
Statistical Analysis 1: Comparison: GEn 1200 mg vs GEn 3600 mg; Test type: Superiority or Other; p = 0.013, ANCOVA; An ANCOVA (repeated measures mixed model) with body mass index, baseline 24-hr average pain intensity, and grouped center as covariates was used; Adjusted mean difference versus placebo = -0.29, 90% CI 2-sided [-0.48 to -0.10]

2. Primary Outcome: Change From Baseline in the Mean 24-hour Average Pain Intensity (API) Score at the Last Week of Each Treatment Period Using LOCF Data for Each Treatment Period
Description: Baseline and end of treatment values are the calculated means of the daily 24-hour API scores for each participant during the last 7 days prior to randomization (baseline) and the last 7 days on treatment within each period (end of treatment). Participants used a hand-held diary to rate their average pain intensity over the preceding 24 hours, using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). LOCF was used if less than 4 days of diary data were provided. The by period summary is provided as a sensitivity analysis for the primary analysis.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, 1 participant did not provide post-baseline data for 24 hour API while taking GEn 3600 mg in the first period, and was therefore not included in this analysis.
Measure: Mean (Standard Deviation); unit: points on a scale
Groups:
- GEn 1200 mg in First Intervention Period: GEn 1200 mg daily in first intervention period only
- GEn 3600 mg in First Intervention Period: GEn 3600 mg daily in first intervention period only
- GEn 1200 mg in Second Intervention Period: GEn 1200 mg daily in second intervention period only
- GEn 3600 mg in Second Interevention Period: GEn 3600 mg daily in second intervention period only
Arm/Group | GEn 1200 mg in First Intervention Period | GEn 3600 mg in First Intervention Period | GEn 1200 mg in Second Intervention Period | GEn 3600 mg in Second Interevention Period
Number analyzed (Participants) | 49 | 43 | 41 | 41
points on a scale | -1.11 (1.477) | -1.09 (1.366) | -1.29 (1.742) | -1.92 (2.000)

3. Secondary Outcome: Change From Baseline in the Mean Day-time Average Pain Intensity (API) Score at the Last Week of Each Treatment Period Using LOCF Data
Description: Day-time is defined as the time between rising in the morning and going to bed at night. Participants recorded day-time API on a daily basis in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and end of treatment scores are as defined for the primary endpoint. Change from baseline is calculated as the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, 1 participant did not provide post-baseline data for day-time pain assessments during the GEn 3600 mg treatment period, and was therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 90 | 84
points on a scale | -1.17 (0.172) | -1.48 (0.174)

4. Secondary Outcome: Change From Baseline in the Mean Day-time Worst Pain Intensity Score at the Last Week of Each Treatment Period Using LOCF Data
Description: Day-time worst pain is defined as the participant's assessment of their worst pain intensity between rising in the morning and going to bed at night. Day-time worst pain was recorded in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and end of treatment scores are as defined for the primary endpoint. Change from baseline is calculated as the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 90 | 84
points on a scale | -1.17 (0.178) | -1.50 (0.181)

5. Secondary Outcome: Change From Baseline in the Mean Current (Evening) Pain Intensity Score at the Last Week of Each Treatment Period Using LOCF Data
Description: Current pain is defined as the participant's assessment of pain intensity "right now." Participants recorded their current evening pain intensity in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and end of treatment scores are as defined for the primary endpoint. Change from baseline is calculated as the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, 1 participant did not provide post-baseline data for current evening pain during the GEn 3600 mg treatment period, and was therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 90 | 84
points on a scale | -1.10 (0.180) | -1.39 (0.183)

6. Secondary Outcome: Change From Baseline in the Mean Night-time Average Pain Intensity (API) Score at the Last Week of Each Treatment Period Using LOCF
Description: Night-time is defined as the time between going to bed in the evening and rising in the morning. Participants recorded night-time API on a daily basis in the morning upon wakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and end of treatment scores are as defined for the primary endpoint. Change from baseline is calculated as the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, 1 participant did not provide post-baseline data for night-time pain assessments during the GEn 1200 mg treatment period, and was therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 89 | 85
points on a scale | -0.92 (0.188) | -1.21 (0.190)

7. Secondary Outcome: Change From Baseline in the Mean Night-time Worst Pain Intensity Score at the Last Week of Each Treatment Period Using LOCF
Description: Night-time worst pain is defined as the participant's assessment of their worst pain intensity between going to bed and rising in the morning. Participants recorded night-time worst pain in the morning upon wakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and end of treatment scores are as defined for primary endpoint. Change from baseline = the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 89 | 85
points on a scale | -0.97 (0.192) | -1.33 (0.194)

8. Secondary Outcome: Change From Baseline in the Mean Current Morning Pain Intensity Score at the Last Week of Each Treatment Period Using LOCF
Description: Current pain is defined as the participant's assessment of pain intensity "right now." Participants recorded their current morning pain intensity in the morning upon wakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and end of treatment scores are as defined for the primary endpoint. Change from baseline is calculated as the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, 1 participant did not provide post-baseline data for current morning pain during the GEn 1200 mg treatment period, and was therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 89 | 85
points on a scale | -1.11 (0.187) | -1.46 (0.189)

9. Secondary Outcome: Number of Participants Achieving Various Levels of Percent Reduction From Baseline in the Mean 24-hour Average Pain Intensity Score at the Last Week of Each Treatment Period Using LOCF Data
Description: Baseline and end of treatment (EOT) scores are the calculated means of the 24-hour average pain scores for each participant during the last 7 days prior to randomization (Baseline) and the 7 days prior to the last on-treatment completed diary (EOT). Percent reduction from baseline was calculated as the [(EOT score minus baseline score) divided by the baseline score], multiplied by 100. The PI-NRS is an 11-point scale (0=no pain, 10=pain as bad as you can imagine) by which a participant assesses their 24-hour average pain intensity. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, there was one participant who did not provide post-baseline data for 24-hour API assessments during the GEn 3600 mg treatment period, and was therefore not included in this analysis.
Measure: Number; unit: participants
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 90 | 84
participants
  0% or more | 68 | 71
  10% or more | 51 | 49
  20% or more | 39 | 42
  30% or more | 28 | 32
  40% or more | 17 | 26
  50% or more | 15 | 16
  60% or more | 6 | 11
  70% or more | 4 | 5
  80% or more | 1 | 2
  90% or more | 1 | 2
  100% | 0 | 2

10. Secondary Outcome: Number of Participants Achieving Various Levels of Percent Reduction From Baseline in the Mean 24-hour Average Pain Intensity Score at the Last Week of Each Treatment Period Using LOCF Data by Period
Description: Baseline and end of treatment scores are the calculated means of the 24-hour average pain scores for each participant during the last 7 days prior to randomization (Baseline) and the 7 days prior to the last on-treatment completed diary (end of treatment). Percent reduction from baseline was calculated as the [(end of treatment score minus the baseline score) divided by the baseline score], multiplied by 100. The PI-NRS is an 11-point scale (0=no pain, 10=pain as bad as you can imagine) by which a participant assesses their 24-hour average pain intensity. Data are summarized by period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, there was one participant who did not provide post-baseline data for 24-hour API while taking GEn 3600 mg in the first period, and was therefore not included in this analysis.
Measure: Number; unit: participants
Groups:
- GEn 1200 mg in First Intervention Period: GEn 1200 mg daily in first intervention period
- GEn 3600 mg in First Intervention Period: GEn 3600 mg daily in first intervention period
- GEn 1200 mg in Second Intervention Period: GEn 1200 mg daily in second intervention period
- GEn 3600 mg in Second Intervention Period: GEn 3600 mg daily in second intervention period
Arm/Group | GEn 1200 mg in First Intervention Period | GEn 3600 mg in First Intervention Period | GEn 1200 mg in Second Intervention Period | GEn 3600 mg in Second Intervention Period
Number analyzed (Participants) | 49 | 43 | 41 | 41
participants
  0% or more | 38 | 34 | 30 | 37
  10% or more | 26 | 23 | 25 | 26
  20% or more | 19 | 19 | 20 | 23
  30% or more | 13 | 13 | 15 | 19
  40% or more | 9 | 10 | 8 | 16
  50% or more | 7 | 5 | 8 | 11
  60% or more | 1 | 3 | 5 | 8
  70% or more | 0 | 0 | 4 | 5
  80% or more | 0 | 0 | 1 | 2
  90% or more | 0 | 0 | 1 | 2
  100% | 0 | 0 | 0 | 2

11. Secondary Outcome: Change From Baseline in the Mean Daily Dose in Milligrams of Rescue Medication at the Last Week of Each Treatment Period
Description: Mean daily use of rescue medication (milligrams of acetaminophen) was calculated by determining the average number of tablets taken per day of rescue medication (Commercial Tylenol) during treatment and multiplying that by 500 mg. Baseline and end of treatment scores are as defined for the primary endpoint. Change from baseline is calculated as the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, there was one participant who did not provide post-baseline data for rescue medication usage during the GEn 3600 mg treatment period, and was therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: milligrams
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 90 | 84
milligrams | -68.18 (73.404) | -71.26 (74.746)

12. Secondary Outcome: Number of Participants Who Are Responders on the Patient Global Impression of Change (PGIC) at the Last Week of Each Treatment Period Using LOCF Data
Description: The PGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the participant's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved" Data are summarized by dose, independent of treatment period.
Time Frame: End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: ITT Population. There were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. There were many participants who did not respond to the questionnaire and thus could not be included in the analysis.
Measure: Number; unit: participants
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 63 | 61
participants | 17 | 28

13. Secondary Outcome: Number of Participants Who Are Responders on the Patient Global Impression of Change (PGIC) Questionnaire at the Last Week of Each Treatment Period Presented by Period Using LOCF Data
Description: The PGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the participant's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved". Data are summarized by dose within each treatment period.
Time Frame: End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: as for outcome 12
Measure: Number; unit: participants
Groups:
- GEn 3600 mg in Second Intervention Period: GEn 3600 mg daily either in second intervention period
Arm/Group | GEn 1200 mg in First Intervention Period | GEn 3600 mg in First Intervention Period | GEn 1200 mg in Second Intervention Period | GEn 3600 mg in Second Intervention Period
Number analyzed (Participants) | 35 | 27 | 28 | 34
participants | 6 | 11 | 11 | 17

14. Secondary Outcome: Number of Participants Who Are Responders on the Clinical Global Impression of Change (CGIC) Questionnaire at the Last Week of Each Treatment Period Using LOCF Data
Description: The CGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the clinician's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved." Data are summarized by dose, independent of treatment period.
Time Frame: End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: ITT Population. There were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. There were many participants without a response to this questionnaire and thus could not be included in the analysis.
Measure: Number; unit: participants
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 53 | 48
participants | 15 | 18

15. Secondary Outcome: Number of Participants Who Are Responders on the Clinical Global Impression of Change (CGIC) Questionnaire at the Last Week of Each Treatment Period Presented by Period Using LOCF Data
Description: The CGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the clinician's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved." Data are summarized by dose within each treatment period.
Time Frame: End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: ITT Population. There were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. There were many participants without a response data to this questionnaire and could thus not be included in the analysis.
Measure: Number; unit: participants
Arm/Group | GEn 1200 mg in First Intervention Period | GEn 3600 mg in First Intervention Period | GEn 1200 mg in Second Intervention Period | GEn 3600 mg in Second Intervention Period
Number analyzed (Participants) | 28 | 22 | 25 | 26
participants | 5 | 8 | 10 | 10

16. Secondary Outcome: Change From Baseline in the Mean Sleep Interference Score at the Last Week of Each Treatment Period Using LOCF Data
Description: Participants assessed sleep interference due to pain on a daily basis using the 11-point NRS (0=pain does not interfere with sleep, 10=pain completely interferes with sleep). Baseline and end of treatment scores are as defined for the primary endpoint. Change from baseline is calculated as the end of treatment score minus the baseline score. An ANCOVA with baseline value, BMI, grouped center as covariates was used. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of each treatment period)
Population: Of the 93 participants in the ITT Population, there were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. In addition, 1 participant did not provide post-baseline data for sleep interference during the GEn 1200 mg treatment period, and was therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 89 | 85
points on a scale | -0.97 (0.205) | -1.23 (0.207)

17. Secondary Outcome: Change From Baseline in the Severity of Pain and the Impact of Pain as Assessed by the Brief Pain Inventory (BPI) at the Last Week of Each Treatment Period Using LOCF
Description: The BPI assesses the severity and interference of pain; and consists of 6 items assessed on an 11-point NRS (0=no impact to 10=greatest impact). 2 summary scores are calculated: BPI Severity Score (average of first 4 items) and BPI Interference Score (average of 7 responses to item 6); where scores range from 0 to 10 (0=no impact to 10=greatest impact). Analysis of this endpoint is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates. Data are summarized by dose, independent of treatment period.
Time Frame: Baseline and End of Treatment (Weeks 4 and 9, representing the last week of treatment)
Population: ITT Population. There were 3 and 8 participants who did not take GEn 1200 and 3600 mg, respectively, in the second period. There were many participants who did not respond to the questionnaire and could thus not be included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | GEn 1200 mg | GEn 3600 mg
Number analyzed (Participants) | 62 | 60
points on a scale
  Brief Pain Inventory Severity of Pain | -1.17 (0.223) | -1.63 (0.225)
  Brief Pain Inventory Interference of Pain | -0.82 (0.244) | -1.57 (0.247)

18. Secondary Outcome: Mean Gabapentin Steady-State (ss) Average, Minimum and Maximum Concentrations
Description: Steady-state average (Cave, ss), maximum (Cmax, ss), and minimum (Cmin,ss) plasma concentration of gabapentin in each participant were estimated using the gabapentin plasma concentration data and with the aid of a population pharmacokinetic model. Dispersion is represented by the fifth to ninety-fifth percentile, though labeled as "Full Range." A total of 10 blood samples were collected per participant over the Baseline, Period 1, and Period 2 at various timepoints during the dosing interval. Plasma concentration of gabapentin in these samples was measured.
Time Frame: A total of 10 blood samples (2 samples at each visit) were collected per participant at Baseline, and the Week 1 and Week 4 visits for each period
Population: Drug concentration data were available from 89 ITT Population participants. Data from 7 of these participants had one concentration with less than half of the first percentile of the concentrations observed at ss and were defined as non-compliant and were excluded from the pharmacokinetic (PK) analysis.
Measure: Geometric Mean (Full Range); unit: micrograms per milliliter
Groups:
- GEn 1200 mg: PK population from GEn 1200 mg treatment daily from either first intervention period or second intervention period
- GEn 3600 mg: PK population from GEn 3600 mg treatment daily from either first intervention period or second intervention period
- Gabapentin 1800 mg: PK population from Gabapentin 1800 mg Baseline Treatment period
Arm/Group | GEn 1200 mg | GEn 3600 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 82 | 82 | 82
micrograms per milliliter
  Cave,ss | 4.1 [2.9 to 7.4] | 12.4 [8.5 to 22.2] | 6.8 [3.8 to 13.4]
  Cmin, ss | 3.0 [1.7 to 6.1] | 9.2 [4.5 to 18.5] | 4.3 [2.3 to 9.4]
  Cmax, ss | 5.1 [3.4 to 9.0] | 15.2 [9.9 to 27.0] | 7.4 [4.3 to 13.7]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the start of the baseline gabapentin treatment period through the post-treatment follow-up visit (up to Week 11).
Description: The AEs reported to start or worsen during the treatment phase of the study are presented.
Groups:
- Baseline Gabapentin 1800 mg: Gabapentin 1800 mg daily for 2 weeks before randomization. Only includes participants who were subsequently randomized.
- Crossover GEn 2400 mg: GEn 2400 mg daily during 4-day crossover period in between the first intervention period and the second intervention period
- Down-Titration Period: Participants down- titrated from GEn 3600 mg/day by taking 2400 mg/day for 2 days, followed by 1200 mg/day for 2 days, followed by 600 mg/day for 2 days before ending the assigned treatment. Participants down- titrated from GEn 1200 mg/day by taking 1200 mg/day for 3 days, followed by 600 mg/day for 3 days before ending the assigned treatment.
- Overall GEn: All participants receiving GEn in any treatment period
Arm/Group | Baseline Gabapentin 1800 mg | GEn 1200 mg | Crossover GEn 2400 mg | GEn 3600 mg | Down-Titration Period | Overall GEn
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/91 | 0/82 | 0/85 | 1/80 | 1/94
Other Adverse Events (participants affected / at risk) | 2/94 | 15/91 | 3/82 | 14/85 | 2/80 | 27/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline Gabapentin 1800 mg (N=94) | GEn 1200 mg (N=91) | Crossover GEn 2400 mg (N=82) | GEn 3600 mg (N=85) | Down-Titration Period (N=80) | Overall GEn (N=94)
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline Gabapentin 1800 mg (N=94) | GEn 1200 mg (N=91) | Crossover GEn 2400 mg (N=82) | GEn 3600 mg (N=85) | Down-Titration Period (N=80) | Overall GEn (N=94)
Nasopharyngitis (Infections and infestations) | 0 | 4 | 0 | 1 | 0 | 5
Headache (Nervous system disorders) | 1 | 1 | 0 | 3 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 3 | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1 | 4
Fatigue (General disorders) | 0 | 0 | 1 | 2 | 0 | 3
Post herpetic neuralgia (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 3
Somnolence (Nervous system disorders) | 0 | 3 | 0 | 2 | 0 | 3
Odema peripheral (General disorders) | 1 | 1 | 0 | 1 | 0 | 2
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 2
Irritability (General disorders) | 0 | 2 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.